CLINICAL TRIAL: NCT00741780
Title: Long-term Observational Follow-up Study of a Multicenter, Randomized, Double-blind, Placebo-controlled, Comparative Trial of AMD3100 (240µg/kg) Plus G-CSF (10µg/kg) Versus G-CSF (10µg/kg) Plus Placebo to Mobilize and Collect ≥ 6X 10^6 CD34+ Cells/kg in Multiple Myeloma Patients for Autologous Transplantation
Brief Title: Long-Term Follow-up Study for Multiple Myeloma Patients Who Received Study Treatment (Plerixafor or Placebo) in the AMD3100-3102 Study (NCT00103662).
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AMD31003102LTF
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma; Autologous Transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — plerixafor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- G-CSF plus plerixafor: Participants in AMD3100-3102 (NCT00103662) who underwent mobilization with granulocyte colony-stimulating factor (G-CSF) and received plerixafor prior to undergoing apheresis.
  Interventions: Drug: plerixafor; Drug: granulocyte colony-stimulating factor (G-CSF)
- G-CSF plus placebo: Participants in AMD3100-3102 (NCT00103662) who underwent mobilization with granulocyte colony-stimulating factor (G-CSF) and received placebo prior to undergoing apheresis.
  Interventions: Drug: Placebo; Drug: granulocyte colony-stimulating factor (G-CSF)

INTERVENTIONS:
Drug: Placebo
  Groups: G-CSF plus placebo
Drug: plerixafor
  Other Names: Mozobil; AMD3100
  Groups: G-CSF plus plerixafor
Drug: granulocyte colony-stimulating factor (G-CSF)

SUMMARY:
This is a long-term observational study of patients that were treated with at least 1 dose of study treatment (plerixafor or placebo) in the AMD3100-3102 protocol (NCT00103662).

DETAILED DESCRIPTION:
This is a long-term observational study of patients who received at least one dose of study treatment (plerixafor or placebo) in a multicenter, randomized, double blind, placebo-controlled study to evaluate AMD3100 plus granulocyte colony stimulating factor (GCSF) versus G-CSF plus placebo to mobilize and transplant Multiple Myeloma (MM) patients (protocol AMD31003102LTF [NCT00103662]). The objective of this study is to assess progression-free survival and overall survival of patients treated with at least 1 dose of study treatment (placebo or plerixafor) for a period of 5 years following the first dose of study treatment (placebo or plerixafor) in protocol AMD3100-3102 (NCT00103662).

ELIGIBILITY:
Inclusion Criteria:

* All patients who received a dose of study treatment (plerixafor or placebo) in protocol AMD3100-3102 (NCT00103662)

Exclusion Criteria:

* No Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the AMD3100-3102 study (NCT00103662) who received a at least one dose of study treatment (plerixafor or placebo).
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2006-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival and overall survival of patients treated with at least 1 dose of study treatment (placebo or plerixafor) in protocol AMD3100-3102 (NCT00103662) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company

REFERENCES:
- [Derived] Micallef IN, Stiff PJ, Nademanee AP, Maziarz RT, Horwitz ME, Stadtmauer EA, Kaufman JL, McCarty JM, Vargo R, Cheverton PD, Struijs M, Bolwell B, DiPersio JF. Plerixafor Plus Granulocyte Colony-Stimulating Factor for Patients with Non-Hodgkin Lymphoma and Multiple Myeloma: Long-Term Follow-Up Report. Biol Blood Marrow Transplant. 2018 Jun;24(6):1187-1195. doi: 10.1016/j.bbmt.2018.01.039. Epub 2018 Feb 2. PMID 29410180